CLINICAL TRIAL: NCT00291642
Title: Double Blind, Double-dummy, Five Parallel Groups, Randomized, Exploratory Clinical Trial to Compare the Efficacy of Single Dose of Levocetirizine 2.5 mg Oral Drops (5 mg/mL), Levocetirizine 5 mg Oral Tablets, Cetirizine 5 mg Oral Drops (10 mg/mL) and Cetirizine 10 mg Oral Tablets to Placebo in Reducing Symptoms of Seasonal Allergic Rhinitis (SAR) in Ragweed Sensitive Subjects Exposed to Ragweed Pollen in an Environmental Exposure Unit (EEU)
Brief Title: A Study to Compare the Efficacy of Levocetirizine to Placebo in Reducing Symptoms of Seasonal Allergic Rhinitis (SAR) in Sensitive Subjects Exposed to Ragweed Pollen
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A00412
Record Dates: First submitted 2006-02-10; First posted 2006-02-14 (Estimated); Results first posted 2018-07-20 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08-01

CONDITIONS: Rhinitis; Allergic; Seasonal
Keywords: Levocetirizine; Xyzal; Rhinitis; Allergic; Seasonal; Ragweed
MeSH Terms: conditions — Rhinitis | interventions — levocetirizine; Cetirizine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (PBO) (Placebo Comparator): A single dose of placebo was administered orally on Day 1.
  Interventions: Drug: Placebo drops; Drug: Placebo tablets matching to levocetirizine; Drug: Placebo tablets matching to cetirizine
- Levocetirizine (LCTZ) 2.5 mg (Experimental): A single dose of 2.5 mg of LCTZ oral drops was administered orally on Day 1.
  Interventions: Drug: Levocetirizine drops
- Levocetirizine (LCTZ) 5 mg (Experimental): A single dose of 5 mg of LCTZ oral tablet was administered orally on Day 1.
  Interventions: Drug: Levocetirizine tablets
- Cetirizine (CTZ) 5 mg (Experimental): A single dose of 5 mg of CTZ oral drops was administered orally on Day 1.
  Interventions: Drug: Cetirizine drops
- Cetirizine (CTZ) 10 mg (Experimental): A single dose of 10 mg of CTZ oral tablet was administered orally on Day 1.
  Interventions: Drug: Cetirizine tablets

INTERVENTIONS:
Drug: Placebo drops — * Pharmaceutical form: Drops for oral administration
  * Route of administration: Oral use
  Arms: Placebo (PBO)
Drug: Placebo tablets matching to levocetirizine — * Pharmaceutical form: Tablets for oral administration
  * Route of administration: Oral use
  Arms: Placebo (PBO)
Drug: Placebo tablets matching to cetirizine — * Pharmaceutical form: Tablets for oral administration
  * Route of administration: Oral use
  Arms: Placebo (PBO)
Drug: Levocetirizine drops — * Pharmaceutical form: Drops for oral administration
  * Concentration: 5 mg/ml
  * Route of administration: Oral use
  Other Names: Xyzal
  Arms: Levocetirizine (LCTZ) 2.5 mg
Drug: Levocetirizine tablets — * Pharmaceutical form: Tablets for oral administration
  * Concentration: 5 mg
  * Route of administration: Oral use
  Other Names: Xyzal
  Arms: Levocetirizine (LCTZ) 5 mg
Drug: Cetirizine drops — * Pharmaceutical form: Drops for oral administration
  * Concentration: 10 mg/ml
  * Route of administration: Oral use
  Arms: Cetirizine (CTZ) 5 mg
Drug: Cetirizine tablets — * Pharmaceutical form: Tablets for oral administration
  * Concentration: 10 mg
  * Route of administration: Oral use
  Arms: Cetirizine (CTZ) 10 mg

SUMMARY:
The purpose of the study is to assess the efficacy comparability of cetirizine and levocetirizine, by comparing the effects of single intake of the two drugs to placebo in reducing symptoms of seasonal allergic rhinitis (SAR) in ragweed sensitive adult subjects exposed to ragweed pollen in an Environmental Exposure Unit.

ELIGIBILITY:
Inclusion Criteria:

* Female subject of non-childbearing potential or of childbearing potential agreeing not to become pregnant during the study.
* Have had seasonal allergic rhinitis due to Ragweed for the last 2 consecutive years
* Subjects who obtain a minimum sum considering SAR related symptoms (mean value) as defined by protocol

Exclusion Criteria:

* Any clinically significant condition that might interfere with the treatment evaluation, both for efficacy and safety
* Have used forbidden concomitant medications as defined by the protocol

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 551 (Actual)
Dates: Start 2006-01-01; Primary Completion 2006-04-01 (Actual); Study Completion 2006-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — UCB (+1 844 599 2273)
Locations (1):
- Kingston, Ontario, Canada

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participant Flow refers to the Randomized Set.
Period: Overall Study
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg
Started | 78 | 116 | 119 | 119 | 119
Completed | 76 | 116 | 117 | 119 | 118
Not Completed | 2 | 0 | 2 | 0 | 1
Not completed — Adverse Event | 1 | 0 | 1 | 0 | 1
Not completed — Patient missed visit | 0 | 0 | 1 | 0 | 0
Not completed — Intake of prohibited medication | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Intention-to-Treat (ITT) Set.
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg | Total Title
Number analyzed (Participants) | 78 | 116 | 119 | 119 | 119 | 551
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 2 | 6 | 4 | 15
  Between 18 and 65 years | 76 | 113 | 114 | 113 | 114 | 530
  >=65 years | 1 | 1 | 3 | 0 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.71 (12.46) | 33.45 (11.28) | 34.36 (12.84) | 32.91 (11.30) | 34.33 (11.65) | 33.76 (11.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 65 | 68 | 65 | 72 | 312
  Male | 36 | 51 | 51 | 54 | 47 | 239

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Major Symptom Complex (MSC) Score Over Period I
Description: Six individual symptoms which are most dominant in the rhinitis symptom profile will be combined to form the MSC severity score:
  Runny nose (right and left), itchy nose (right and left), sniffles, nose blows, sneezes, watery eyes.
  Each individual symptom, except nose blows and sneezes, is rated on a 5-point scale of severity: 0 = None, 1 = a little, 2 = Moderate, 3 = Quite a bit, 4 = severe, 5 = very severe. For nose blows and sneezes, the subjects had to record the number of each symptom since last evaluation. This number corresponds to a score ranging from 0 to 8. The total MSC score ranges from 0 - 36. Increasing scores are associated with increasing severity. Negative values indicate improvement from Baseline.
Time Frame: Baseline, Treatment Period 1 [Day 1, from drug intake (at 11:00 am) to 5 hours post-treatment (at 4:00 pm)]
Population: Only patients with valid MSC scores in Period I were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg
Number analyzed (Participants) | 78 | 116 | 119 | 119 | 119
units on a scale | -3.80 (0.495) | -7.15 (0.406) | -7.05 (0.401) | -7.93 (0.401) | -7.54 (0.401)
Statistical Analysis 1: Comparison: Placebo (PBO) vs Levocetirizine (LCTZ) 2.5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -3.35, 95% CI 2-sided [-4.61 to -2.09], Standard Error of Mean 0.640
Statistical Analysis 2: Comparison: Placebo (PBO) vs Levocetirizine (LCTZ) 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -3.25, 95% CI 2-sided [-4.50 to -2.00], Standard Error of Mean 0.637
Statistical Analysis 3: Comparison: Placebo (PBO) vs Cetirizine (CTZ) 5 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -4.13, 95% CI 2-sided [-5.38 to -2.88], Standard Error of Mean 0.637
Statistical Analysis 4: Comparison: Placebo (PBO) vs Cetirizine (CTZ) 10 mg; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -3.74, 95% CI 2-sided [-4.99 to -2.49], Standard Error of Mean 0.637

2. Secondary Outcome: Change From Baseline in the MSC Score Over Period II
Description: as for outcome 1
Time Frame: Baseline, Treatment Period II [Day 2, (8:30 am to 12:00 pm)]
Population: Only patients with valid MSC scores in Period II were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg
Number analyzed (Participants) | 76 | 116 | 117 | 119 | 118
units on a scale | -3.50 (0.604) | -6.35 (0.489) | -7.07 (0.487) | -6.78 (0.483) | -7.92 (0.485)

3. Secondary Outcome: Change From Baseline in the MSC Score Over the Total Treatment Period (Period I + Period II)
Description: as for outcome 1
Time Frame: Baseline to Day 2
Population: Only patients with valid MSC scores in Period I and II were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg
Number analyzed (Participants) | 78 | 116 | 119 | 119 | 119
units on a scale | -3.61 (0.473) | -6.80 (0.388) | -7.10 (0.383) | -7.43 (0.384) | -7.72 (0.383)

4. Secondary Outcome: Change From Baseline in the Total Symptom Complex (TSC) Score Over Period I
Description: The TSC score was calculated as the sum of the following 10 individual symptom scores:
  runny nose (left and right), itchy nose (left and right), sniffles, nose blows, sneezes, watery eyes, itchy eyes and ears, itchy throat, cough and postnasal drip.
  Each individual symptom, except nose blows and sneezes, is rated on a 5-point scale of severity: 0 = None, 1 = a little, 2 = Moderate, 3 = Quite a bit, 4 = severe, 5 = very severe. For nose blows and sneezes, the subjects had to record the number of each symptom since last evaluation. This number corresponds to a score ranging from 0 to 8. The TSC score ranges from 0 to 56. Increasing scores are associated with increasing severity. Negative values indicate improvement from Baseline.
Time Frame: Baseline, Treatment Period I [Day 1, from drug intake (at 11:00 am) to 5 hours post-treatment (at 4:00 pm)]
Population: Only patients with valid TSC scores in Period I were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg
Number analyzed (Participants) | 78 | 116 | 119 | 119 | 119
units on a scale | -6.55 (0.757) | -11.33 (0.620) | -11.27 (0.613) | -12.71 (0.613) | -11.74 (0.613)

5. Secondary Outcome: Change From Baseline in the Total Symptom Complex (TSC) Score Over Period II
Description: as for outcome 4
Time Frame: Baseline, Treatment Period II [Day 2, (8:30 am to 12:00 pm)]
Population: Only patients with valid TSC scores in Period II were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg
Number analyzed (Participants) | 76 | 116 | 117 | 119 | 118
units on a scale | -5.73 (0.917) | -10.25 (0.742) | -11.03 (0.739) | -10.73 (0.734) | -12.14 (0.736)

6. Secondary Outcome: Change From Baseline in the Total Symptom Complex (TSC) Score Over the Total Treatment Period (Period I + Period II)
Description: as for outcome 4
Time Frame: Baseline to Day 2
Population: Only patients with valid TSC scores in Period I and II were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg
Number analyzed (Participants) | 78 | 116 | 119 | 119 | 119
units on a scale | -6.10 (0.729) | -10.86 (0.598) | -11.22 (0.591) | -11.84 (0.591) | -11.92 (0.591)

7. Secondary Outcome: Change From Baseline in the Individual Symptom Scores Over Period I
Description: Individual symptom scores include Runny Nose Score, Itchy Nose Score, Sniffles Score, Watery Eyes Score, Sneezes Score, Nose Blows Score.
  The subjects had to evaluate the severity of the symptoms using a scale from "None" to "Very severe" (ranging from 0 to 5).
  For Sneezes Score and Nose Blows Score, the subjects had to record the number of each symptom since last evaluation. This number corresponds to a score ranging from 0 to 8.
  Increasing scores are associated with increasing severity. Negative values indicate improvement from Baseline.
Time Frame: Baseline, Treatment Period 1 [Day 1, from drug intake (at 11:00 am) to 5 hours post-treatment (at 4:00 pm)]
Population: Only subjects with valid individual symptom scores in Period I were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg
Number analyzed (Participants) | 78 | 116 | 119 | 119 | 119
units on a scale
  Runny Nose Score | -0.60 (0.095) | -1.01 (0.078) | -0.95 (0.077) | -1.17 (0.077) | -1.04 (0.077)
  Itchy Nose Score | -0.66 (0.099) | -1.03 (0.082) | -1.09 (0.081) | -1.28 (0.081) | -1.10 (0.081)
  Sniffles Score | -0.65 (0.100) | -1.15 (0.082) | -1.06 (0.081) | -1.24 (0.081) | -1.10 (0.081)
  Nose Blow Score | -0.98 (0.129) | -1.87 (0.106) | -1.82 (0.105) | -1.92 (0.105) | -1.96 (0.105)
  Sneezes Score | -0.37 (0.103) | -1.15 (0.084) | -1.07 (0.083) | -1.22 (0.083) | -1.23 (0.083)
  Watery Eyes Score | -0.56 (0.090) | -0.94 (0.074) | -1.08 (0.073) | -1.13 (0.073) | -1.07 (0.073)

8. Secondary Outcome: Change From Baseline in the Individual Symptom Scores Over Period II
Description: as for outcome 7
Time Frame: Baseline, Treatment Period II [Day 2, (8:30 am to 12:00 pm)]
Population: Only subjects with valid individual symptom scores in Period II were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg
Number analyzed (Participants) | 76 | 116 | 117 | 119 | 118
units on a scale
  Runny Nose Score | -0.62 (0.122) | -0.86 (0.098) | -0.94 (0.098) | -0.95 (0.097) | -1.10 (0.098)
  Itchy Nose Score | -0.57 (0.120) | -1.00 (0.097) | -1.11 (0.097) | -1.13 (0.096) | -1.24 (0.096)
  Sniffles Score | -0.58 (0.127) | -0.91 (0.103) | -0.96 (0.102) | -0.90 (0.101) | -1.21 (0.102)
  Nose Blow Score | -1.00 (0.162) | -1.61 (0.131) | -1.84 (0.131) | -1.78 (0.130) | -2.02 (0.130)
  Sneezes Score | -0.48 (0.112) | -1.18 (0.091) | -1.33 (0.090) | -1.19 (0.089) | -1.38 (0.090)
  Watery Eyes Score | -0.30 (0.119) | -0.78 (0.097) | -0.91 (0.096) | -0.83 (0.096) | -0.93 (0.096)

9. Secondary Outcome: Change From Baseline in the Individual Symptom Scores Over the Total Treatment Period (Period I + Period II)
Description: as for outcome 7
Time Frame: Baseline to Day 2
Population: Only subjects with valid individual symptom scores in Period I and II were included in the analysis.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg
Number analyzed (Participants) | 78 | 116 | 119 | 119 | 119
units on a scale
  Runny Nose Score | -0.59 (0.093) | -0.94 (0.076) | -0.95 (0.075) | -1.07 (0.075) | -1.06 (0.075)
  Itchy Nose Score | -0.61 (0.097) | -1.02 (0.080) | -1.10 (0.079) | -1.21 (0.079) | -1.16 (0.079)
  Sniffles Score | -0.60 (0.098) | -1.05 (0.080) | -1.02 (0.079) | -1.09 (0.079) | -1.15 (0.079)
  Nose Blow Score | -0.98 (0.124) | -1.75 (0.102) | -1.83 (0.100) | -1.86 (0.101) | -1.99 (0.100)
  Sneezes Score | -0.41 (0.090) | -1.17 (0.074) | -1.19 (0.073) | -1.21 (0.073) | -1.31 (0.073)
  Watery Eyes Score | -0.44 (0.089) | -0.87 (0.073) | -1.01 (0.072) | -1.00 (0.073) | -1.01 (0.072)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Day 1 until up to 9 days after the study drug intake.
Description: Adverse Events refer to the Safety Population consisting of all subjects who were dispensed medication.
Arm/Group | Placebo (PBO) | Levocetirizine (LCTZ) 2.5 mg | Levocetirizine (LCTZ) 5 mg | Cetirizine (CTZ) 5 mg | Cetirizine (CTZ) 10 mg
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/116 | 0/119 | 0/119 | 0/119
Serious Adverse Events (participants affected / at risk) | 0/78 | 0/116 | 0/119 | 0/119 | 0/119
Other Adverse Events (participants affected / at risk) | 5/78 | 10/116 | 9/119 | 13/119 | 7/119
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (PBO) (N=78) | Levocetirizine (LCTZ) 2.5 mg (N=116) | Levocetirizine (LCTZ) 5 mg (N=119) | Cetirizine (CTZ) 5 mg (N=119) | Cetirizine (CTZ) 10 mg (N=119)
Palpitations (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 2 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 1 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Defaecation urgency (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 3 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 2 | 0 | 1 | 2
Paraesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 1 | 1 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 0
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Nasal mucosal disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days